CLINICAL TRIAL: NCT01408368
Title: Five-year Follow up of a Randomized Clinical Trial of Bilateral Subtotal Thyroidectomy Versus Total Thyroidectomy for Graves' Disease.
Brief Title: Subtotal Versus Total Thyroidectomy for Graves' Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Piotr Laidler / Head of the Biomedical Research Committee of the Jagiellonian University, Biomedical Research Committee of the Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBN/501/ZKL/67/L
Record Dates: First submitted 2011-08-02; First posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Thyroid; Goiter
Keywords: Graves' disease; total thyroidectomy; bilateral subtotal thyroidectomy; Graves' ophthalmopathy; morbidity rate
MeSH Terms: conditions — Thyroid Diseases; Goiter; Graves Disease; Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilateral subtotal thyroidectomy (Active Comparator)
  Interventions: Procedure: Bilateral subtotal thyroidectomy
- Total thyroidectomy (Experimental)
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Procedure: Bilateral subtotal thyroidectomy — The intervention consisted of bilateral subtotal thyroidectomy (leaving on both sides of the neck thyroid stumps of approximately 2 g of normal remnant tissue each).
  Other Names: BST
  Arms: Bilateral subtotal thyroidectomy
Procedure: Total thyroidectomy — The intervention consisted of total extracapsular thyroidectomy.
  Other Names: TT
  Arms: Total thyroidectomy

SUMMARY:
The extent of thyroid resection in Graves' disease remains controversial. The aim of this study was to evaluate long-term results of bilateral subtotal thyroidectomy versus total thyroidectomy in patients with Graves' ophthalmopathy.

DETAILED DESCRIPTION:
Graves' disease was first described in 1835. It is an autoimmune disorder caused by antibodies which bind to thyroid-stimulating hormone (TSH) receptors on the thyroid cell membrane. The overt clinical manifestation of this disease is usually characterised by presence of hyperthyroidism, thyroid associated ophthalmopathy and thyroid dermopathy.

Treatment alternatives of Graves' disease include antithyroid medication, radioiodine therapy or thyroidectomy. The antithyroid medication is often used as the initial treatment for patients with newly diagnosed Graves disease in much of the world including Europe, Japan and South America. However, the use of radioiodine is the most common first-line treatment modality in the United States. Thyroidectomy should be considered in special circumstances such as in children and young adults, pregnant women, in the setting of ophthalmopathy, in the presence of thyroid nodules or big goitre, particularly when compressive symptoms, or substernal thyroid extension is diagnosed, as well as in cases of failed hyperthyroidism remission after antithyroid medication in patients refusing possible radioiodine treatment.

The surgical management of Graves' disease remains controversial. Some authors support total thyroidectomy while others prefer various subtotal procedures. Most low-volume surgeons avoid performing total thyroidectomies for Graves' disease owing to the assumed higher complication rates. On the other hand, an increasing number of total thyroidectomies are currently performed in high-volume endocrine surgery units, and the indications for this procedure include not only high-risk thyroid cancer, but also Graves's disease and multinodular goiter. It has been shown that total thyroidectomy for Graves' disease lowers to almost zero the disease recurrence rate. However, other issues like unclear benefit for natural course of Graves' ophthalmopathy balanced against assumed higher risk of morbidity following more radical thyroid resections need to be clarified.

We hypothesized that total thyroidectomy is superior to bilateral subtotal thyroidectomy for long-term control of Graves' disease. The aim of this study was to evaluate long-term results of bilateral subtotal thyroidectomy versus total thyroidectomy in patients with mild and active Graves' ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

* planned thyroid surgery for clinically, biochemically and immunologically diagnosed Graves' disease in patients with mild active ophthalmopathy and the posterior aspects of both thyroid lobes appearing normal on ultrasound of the neck.

Exclusion Criteria:

* previous thyroid or parathyroid surgery,
* recurrent hyperthyroidism after radioiodine ablation,
* history of Graves' disease longer than 24 months,
* thyroid nodules within the posterior aspect/s of thyroid lobe/s,
* suspicion of thyroid cancer,
* inactive Graves' ophthalmopathy,
* moderate to severe active Graves' ophthalmopathy,
* preoperative recurrent laryngeal nerve palsy,
* pregnancy or lactation,
* age < 18 years, or > 65 years,
* ASA 4 grade (American Society of Anaesthesiology),
* inability to comply with the follow-up protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2000-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Long-term control of Graves' disease | up to 60 months postoperatively
  Recurrence rate of hyperthyroidism and change in Graves' ophthalmopathy

SECONDARY OUTCOMES:
Morbidity rate | up to 12 months postoperatively
  recurrent laryngeal nerve injury and hypoparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University, College of Medicine, Department of Endocrine Surgery, 3rd Chair of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Barczynski M, Konturek A, Hubalewska-Dydejczyk A, Golkowski F, Cichon S, Nowak W. Five-year follow-up of a randomized clinical trial of total thyroidectomy versus Dunhill operation versus bilateral subtotal thyroidectomy for multinodular nontoxic goiter. World J Surg. 2010 Jun;34(6):1203-13. doi: 10.1007/s00268-010-0491-7. PMID 20174803
- [Background] Stalberg P, Svensson A, Hessman O, Akerstrom G, Hellman P. Surgical treatment of Graves' disease: evidence-based approach. World J Surg. 2008 Jul;32(7):1269-77. doi: 10.1007/s00268-008-9497-9. PMID 18327526
- [Background] Bartalena L. The dilemma of how to manage Graves' hyperthyroidism in patients with associated orbitopathy. J Clin Endocrinol Metab. 2011 Mar;96(3):592-9. doi: 10.1210/jc.2010-2329. Epub 2010 Dec 29. PMID 21190983
- [Background] Wilhelm SM, McHenry CR. Total thyroidectomy is superior to subtotal thyroidectomy for management of Graves' disease in the United States. World J Surg. 2010 Jun;34(6):1261-4. doi: 10.1007/s00268-009-0337-3. PMID 20033406
- [Background] Barakate MS, Agarwal G, Reeve TS, Barraclough B, Robinson B, Delbridge LW. Total thyroidectomy is now the preferred option for the surgical management of Graves' disease. ANZ J Surg. 2002 May;72(5):321-4. doi: 10.1046/j.1445-2197.2002.02400.x. PMID 12028087
- [Background] Chi SY, Hsei KC, Sheen-Chen SM, Chou FF. A prospective randomized comparison of bilateral subtotal thyroidectomy versus unilateral total and contralateral subtotal thyroidectomy for graves' disease. World J Surg. 2005 Feb;29(2):160-3. doi: 10.1007/s00268-004-7529-7. Epub 2005 Jan 18. PMID 15650802
- [Background] Witte J, Goretzki PE, Dotzenrath C, Simon D, Felis P, Neubauer M, Roher HD. Surgery for Graves' disease: total versus subtotal thyroidectomy-results of a prospective randomized trial. World J Surg. 2000 Nov;24(11):1303-11. doi: 10.1007/s002680010216. PMID 11038198
- [Derived] Barczynski M, Konturek A, Hubalewska-Dydejczyk A, Golkowski F, Nowak W. Randomized clinical trial of bilateral subtotal thyroidectomy versus total thyroidectomy for Graves' disease with a 5-year follow-up. Br J Surg. 2012 Apr;99(4):515-22. doi: 10.1002/bjs.8660. Epub 2012 Jan 27. PMID 22287122